CLINICAL TRIAL: NCT01433380
Title: Phase 1 Study To Evaluate The Effect Of Single Doses Of Pf-05175157 On Pharmacodynamic And Metabolic Parameters In Healthy Volunteers
Brief Title: A Study To Evaluate PF-05175157 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B1731004
Record Dates: First submitted 2011-08-23; First posted 2011-09-13 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Phase 1; Single Doses; Pharmacodynamics; Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 600 mg PF-05175157 (Experimental): Subjects will receive one dose of PF-05175157. The sequence of receiving 600 mg PF-05175157 or placebo will be randomized.
  Interventions: Drug: PF-05175157
- Placebo (Placebo Comparator): Subjects will receive one dose of placebo. The sequence of receiving placebo or 600 mg PF-05175157 will be randomized.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-05175157 — One single dose of PF-05175157 will be administered as a powder-in-capsule in the fasting state in the AM.
  Arms: 600 mg PF-05175157
Drug: Placebo — One single dose of placebo will be administered as a powder-in-capsule in the fasting state in the AM.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the pharmacodynamics of single oral doses of PF-05175157 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.
* Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests.
* In addition, subjects must have normal pulmonary function tests and normal ocular examination.
* Body Mass Index of 20.0 35.0 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Evidence or history of any chronic ongoing or current pulmonary disease.
* History of smoking in the past 5 years or history or evidence of habitual use of other (non smoked) tobacco or nicotine-containing products within 3 months of Screening or positive cotinine test at Screening or Day 0.
* Active ocular disease including infection, glaucoma, seasonal allergies, dry eye symptoms or retinal/optic nerve disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Changes in carbohydrate and lipid metabolism | 24 hours

SECONDARY OUTCOMES:
Pharmacokinetics: 0.5, 1, 1.5, 2.5, 6.5, 10.5, 24 hrs after dosing, parameters: Cmax, Tmax and Area under the Curve (AUC) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Baton Rouge, Louisiana, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1731004&StudyName=A%20Study%20To%20Evaluate%20PF-05175157%20In%20Healthy%20Volunteers